CLINICAL TRIAL: NCT01528176
Title: Vitamin D Metabolism in Chronic Kidney Disease Patients With Vitamin D Deficiency Treated With Cholecalciferol
Brief Title: Vitamin D Metabolism in Chronic Kidney Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Memphis VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, HALA M ALSHAYEB, Principal Investigator, Memphis VA Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 00703; Department of Vetrans Affair (Other: Department of Vetrans Affairs)
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Vitamin D Metabolism is in Chronic Kidney Disease
Keywords: FGF-23, CKD, Cyp24, 24,25(OH)2D, vitamin D metabolism
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- (CKD) stages III-V and non -CKD patients (Other): We recruited patients with wide range of eGFR
  Interventions: Drug: 10,000 IU of cholecalciferol for a total of 8 weeks

INTERVENTIONS:
Drug: 10,000 IU of cholecalciferol for a total of 8 weeks — Subjects were treated with weekly oral administration of 10,000 IU of cholecalciferol for a total of 8 weeks in order to correct the vitamin D deficiency.

SUMMARY:
To determine whether or not chronic kidney disease (CKD), stages III-V and ESRD , is associated with altered vitamin D metabolism related to fibroblast growth factor-23 (FGF-23) stimulation of Cyp24 and whether they have resistance to elevations of 25 Hydroxyvitamin D (25(OH)D3) after cholecalciferol supplementation.

To determine if such resistance is related to enhanced catabolism of (25(OH)related to elevated levels of FGF-23.

DETAILED DESCRIPTION:
1. Patients in the Memphis VA Medical Center with documented vitamin D deficiency, determined by measurements of 25(OH)D3, were recruited for this study. 25(OH)D3 measurements are commonly obtained during routine clinical care in both primary care and nephrology clinics. Patient with a wide range of kidney function, ranging from normal estimated glomerular filtration rate (e GFR) to patients with stage III and V (CKD) (estimated GFR <60 ml/min) were recruited treated with weekly oral administration of 10,000 IU of cholecalciferol for a total of 8 weeks in order to correct the vitamin D deficiency.
2. Data collected:

   Baseline characteristics including demographics, laboratory data obtained at primary care clinic visits, clinical data from the VAMC medical record and medications were obtained at the time of inclusion into the study. Serum concentrations of FGF23, 25(OH)D, 1,25 dihydroxyvitamin D(1,25 (OH)₂D), 24,25 dihydroxyvitamin D(24,25(OH)₂D) ,intact parathyroid hormone (PTH), Calcium, Phosphorous and creatinine and urinary concentrations of calcium, phosphate and creatinine from 24 hr urine collections were obtained at the time of inclusion into the study and after 8 weeks of weekly cholecalciferol therapy. Serum and buffy coats which were recollected from dialysis patient's who agreed to participate, were used to measure mRNA levels of FGF-23, CPY27B1 and Cyp 24 expression.
3. Methods utilized in analyzing and interpreting the data Descriptive statistics will be performed to compare serum and urinary measurements before and after cholecalciferol therapy. Associations between estimated glomerular filtration rate and levels of vitamin D metabolites and FGF23, before and after treatment, will also be evaluated. The mRNA expression of FGF-23, CPY27B1 and Cyp 24 will be measured in a subset of dialysis patients who completed the treatment course and agreed to provide the additional samples.
4. Duration of the project: 1 year.

ELIGIBILITY:
Inclusion Criteria:

* age 18-85 years; CKD stage III or V; serum 25(OH)D level ≤ 30ng/ml, and serum PTH levels > 70 pg/ml within the last 6 months, informed Consent.

Exclusion Criteria:

* A history of liver disease, sarcoidosis, intestinal malabsorption;
* requirement of dialysis during the study; serum calcium level >10.5 mg/dl,
* calcium-phosphorus product > 70, or
* calcimimetics, or
* phosphorus binders; or
* medications that could affect vitamin D metabolism or
* history of parathyroidectomy.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Vitamin D Metabolism in CKD and ESRD Patients with Vitamin D Deficiency treated with Cholicalciferol | 8 weeks
  Measuring 25(OH)D, FGF23, 24,25(OH)₂D, and 1,25(OH)₂D , PTH, Calcium, Phosphorus at baseline and after 8 weeks of cholecalciferol in a cohort of patients with CKD and non CKD who were having vitamin D defeciency treated with cholecalciferol for 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barry M Wall, MD, Principal Investigator — Memphis , TN ,VAMC; HALA M Alshayeb, MD, Principal Investigator — UTHSC, UCH
Locations (1):
- Memphis Veteran Affair Medical center, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Alshayeb H, Showkat A, Wall BM, Gyamlani GG, David V, Quarles LD. Activation of FGF-23 mediated vitamin D degradative pathways by cholecalciferol. J Clin Endocrinol Metab. 2014 Oct;99(10):E1830-7. doi: 10.1210/jc.2014-1308. Epub 2014 Jun 24. PMID 24960544